CLINICAL TRIAL: NCT01524783
Title: A Randomized, Double-blind, Multicenter, Phase III Study of Everolimus (RAD001) Plus Best Supportive Care Versus Placebo Plus Best Supportive Care in the Treatment of Patients With Advanced NET of GI or Lung Origin
Brief Title: Everolimus Plus Best Supportive Care vs Placebo Plus Best Supportive Care in the Treatment of Patients With Advanced Neuroendocrine Tumors (GI or Lung Origin)
Acronym: RADIANT-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001T2302; 2011-002887-26 (Registry Identifier: EudraCT)
Record Dates: First submitted 2011-12-22; First posted 2012-02-02 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Advanced NET of GI Origin; Advanced NET of Lung Origin; Neuroendocrine Tumors
Keywords: Neuroendocrine tumor; NET; progressive; advanced; gastrointestinal; GI or lung origin; nonfunctional; everolimus; Advanced NET of GI origin; Advanced NET of lung origin
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Everolimus + BSC (Experimental): Participants received everolimus 10 mg once daily plus best supportive care (BSC) throughout the study
  Interventions: Drug: Everolimus; Other: Best suportive care (BSC)
- Placebo + BSC (Placebo Comparator): Participants received matching placebo once daily plus best supportive care (BSC) during the blinded period. Participants were allowed to crossover to treatment with everolimus 10mg once daily plus BSC during the open-label period.
  Interventions: Drug: Placebo; Other: Best suportive care (BSC)

INTERVENTIONS:
Drug: Everolimus — Participants were treated with everolimus 10 mg (two 5 mg tablets) once daily orally taken
  Other Names: RAD001
  Arms: Everolimus + BSC
Drug: Placebo — Participants were treated with two tablets of matching placebo once daily orally taken.
  Arms: Placebo + BSC
Other: Best suportive care (BSC) — Best supportive care includes all care provided to participants deemed necessary by the treating physician, such as but not restricted to anti-diarrheals and analgesics. The optimal care of the patient is based on the treating physician's best medical judgment.

SUMMARY:
The purpose of this study is to compare the antitumor activity of everolimus plus best supportive care versus placebo plus best supportive care in patients with progressive nonfunctional neuroendocrine tumor (NET) of gastrointestinal (GI) or lung origin without a history of, or current symptoms of carcinoid syndrome.

DETAILED DESCRIPTION:
This was a prospective, multi-center, randomized, double-blind, parallel-group, placebo-controlled, two-arm Phase III study comparing the efficacy and safety of everolimus 10 mg daily to placebo in patients with advanced NET of GI or lung origin without a history of, or current symptoms of carcinoid syndrome.

After assessment of eligibility, participants qualifying for the study were randomized in a 2:1 ratio to receive either everolimus or matching placebo. Participants received daily oral doses of 10 mg everolimus or matching placebo as study drug. In both arms, the study drug was combined with best supportive care and treatment cycles were defined as 28 days. Participants were treated until disease progression as per Response Evaluation Criteria In Solid Tumors (RECIST) 1.0, intolerable toxicity, death, lost to follow-up or consent withdrawal. Regardless of the reason for study drug discontinuation, participants had a safety follow-up visit scheduled 30 days after the last dose of the study drug.

Per data monitoring committee recommendation, all participants on treatment with placebo were allowed to crossover to open-label treatment with everolimus. This change was implemented through protocol amendment 3 (issued on 06-May-2016) after which remaining participants entered into open-label phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, well differentiated (G1 or G2), advanced (unresectable or metastatic), neuroendocrine tumor of GI or lung origin
* No history of and no active symptoms related to carcinoid syndrome
* In addition to treatment-naive patients, patients previously treated with SSA, Interferon (IFN), one prior line of chemotherapy, and/or PRRT were allowed into the study. Pretreated patients had to have progressed on or after the last treatment
* Radiological documented disease progression within 6 months prior to randomization
* Measurable disease
* WHO performance status ≤1
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Patients with poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, pancreatic islet cell carcinoma, insulinoma, glucagonoma, gastrinoma, goblet cell carcinoid, large cell neuroendocrine carcinoma and small cell carcinoma
* Patients with pancreatic NET or NET of origins other than GI or Lung
* Patients with history of or active symptoms of carcinoid syndrome (e.g. flushing, diarrhea)
* Patients with more than one line of prior chemotherapy
* Prior targeted therapy
* Hepatic intra-arterial embolization within the last 6 months. Cryoablation or radiofrequency ablation of hepatic metastases within 2 months of randomization
* Prior therapy with mTOR inhibitors (e.g. sirolimus, temsirolimus, deforolimus)
* Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus)
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus
* Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy
* Patients who had any severe and/or uncontrolled medical conditions such as:

  * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to randomization, serious uncontrolled cardiac arrhythmia
  * active or uncontrolled severe infection
  * liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA)
* Chronic treatment with corticosteroids or other immunosuppressive agents
* Known history of HIV seropositivity
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria might apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2014-11-28 (Actual); Study Completion 2020-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (87):
- United States (17):
  - University of California San Diego - Moores Cancer Center Regulatory, La Jolla, California
  - Scripps Clinic Regulatory, La Jolla, California
  - Cedars Sinai Medical Center SC, Los Angeles, California
  - University of Colorado Cancer Centre SC, Aurora, Colorado
  - H Lee Moffitt Cancer Center and Research Institute HLM, Tampa, Florida
  - University of Chicago UC SC, Chicago, Illinois
  - Goshen Center for Cancer Care IU Health SC, Indianapolis, Indiana
  - Dana Farber Cancer Institute SC, Boston, Massachusetts
  - Memorial Sloan Kettering MSkCC SC, New York, New York
  - Montefiore Medical Center MMC, The Bronx, New York
  - Oregon Health and Science University OH&SU, Portland, Oregon
  - Vanderbilt University Medical Center Vanderbilt Med Ctr, Nashville, Tennessee
  - Texas Oncology P A Texas Oncology Amarillo, Dallas, Texas
  - Texas Oncology P A TX Oncology Baylor, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center UT MD Anderson Cancer Ctr, Houston, Texas
  - University of Wisconsin / Paul P. Carbone Comp Cancer Center Univ Wisc, Madison, Wisconsin
- Austria (2):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Vienna
- Belgium (4):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Canada (7):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- China (2):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Beijing
- Novartis Investigative Site, Bogotá, Cundinamarca, Colombia
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Germany (7):
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Athens, Greece
- Novartis Investigative Site, Budapest, Hungary
- Italy (10):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Viagrande, CT
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
- Japan (3):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
- Novartis Investigative Site, Amsterdam, Netherlands
- Poland (2):
  - Novartis Investigative Site, Gliwice, Silesian Voivodeship
  - Novartis Investigative Site, Poznan
- Novartis Investigative Site, Rostov-on-Don, Russia
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Bratislava, Slovak Republic, Slovakia
- Novartis Investigative Site, Parktown, South Africa
- South Korea (3):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Spain (3):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
- Taiwan (5):
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Kuei-Shan Chiang, Taoyuan/ Taiwan ROC
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok, THA
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Istanbul
- United Kingdom (5):
  - Novartis Investigative Site, Glasgow, Scotland
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Chan DL, Yao JC, Carnaghi C, Buzzoni R, Herbst F, Ridolfi A, Strosberg J, Kulke MH, Pavel M, Singh S. Markers of Systemic Inflammation in Neuroendocrine Tumors: A Pooled Analysis of the RADIANT-3 and RADIANT-4 Studies. Pancreas. 2021 Feb 1;50(2):130-137. doi: 10.1097/MPA.0000000000001745. PMID 33560090
- [Derived] Buzzoni R, Carnaghi C, Strosberg J, Fazio N, Singh S, Herbst F, Ridolfi A, Pavel ME, Wolin EM, Valle JW, Oh DY, Yao JC, Pommier R. Impact of prior therapies on everolimus activity: an exploratory analysis of RADIANT-4. Onco Targets Ther. 2017 Oct 16;10:5013-5030. doi: 10.2147/OTT.S142087. eCollection 2017. PMID 29081664
- [Derived] Fazio N, Buzzoni R, Delle Fave G, Tesselaar ME, Wolin E, Van Cutsem E, Tomassetti P, Strosberg J, Voi M, Bubuteishvili-Pacaud L, Ridolfi A, Herbst F, Tomasek J, Singh S, Pavel M, Kulke MH, Valle JW, Yao JC. Everolimus in advanced, progressive, well-differentiated, non-functional neuroendocrine tumors: RADIANT-4 lung subgroup analysis. Cancer Sci. 2018 Jan;109(1):174-181. doi: 10.1111/cas.13427. Epub 2017 Nov 9. PMID 29055056
- [Derived] Pavel ME, Singh S, Strosberg JR, Bubuteishvili-Pacaud L, Degtyarev E, Neary MP, Carnaghi C, Tomasek J, Wolin E, Raderer M, Lahner H, Valle JW, Pommier R, Van Cutsem E, Tesselaar MET, Fave GD, Buzzoni R, Hunger M, Eriksson J, Cella D, Ricci JF, Fazio N, Kulke MH, Yao JC. Health-related quality of life for everolimus versus placebo in patients with advanced, non-functional, well-differentiated gastrointestinal or lung neuroendocrine tumours (RADIANT-4): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2017 Oct;18(10):1411-1422. doi: 10.1016/S1470-2045(17)30471-0. Epub 2017 Aug 30. PMID 28838862
- [Derived] Yao JC, Fazio N, Singh S, Buzzoni R, Carnaghi C, Wolin E, Tomasek J, Raderer M, Lahner H, Voi M, Pacaud LB, Rouyrre N, Sachs C, Valle JW, Fave GD, Van Cutsem E, Tesselaar M, Shimada Y, Oh DY, Strosberg J, Kulke MH, Pavel ME; RAD001 in Advanced Neuroendocrine Tumours, Fourth Trial (RADIANT-4) Study Group. Everolimus for the treatment of advanced, non-functional neuroendocrine tumours of the lung or gastrointestinal tract (RADIANT-4): a randomised, placebo-controlled, phase 3 study. Lancet. 2016 Mar 5;387(10022):968-977. doi: 10.1016/S0140-6736(15)00817-X. Epub 2015 Dec 17. PMID 26703889

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At baseline, participants were randomized to either everolimus+BSC or placebo+BSC arm. Two patients randomized to the everolimus arm were not treated due to withdrawal of consent and protocol deviation.
  As per Data Monitoring Committee recommendation (03-Jun-2015), implemented through protocol amendment 3 (issued on 06-May-2016), remaining participants entered the open-label part of the study, where participants in the placebo arm were allowed to crossover to open-label treatment with everolimus
Groups:
- Everolimus + BSC (Throughout Study): Participants received everolimus 10 mg once daily BSC throughout the study
- Placebo+BSC (Blinded Period): Participants received matching placebo once daily plus BSC during the blinded period
- Everolimus+BSC (Crossover): Participants who crossed over from placebo arm (blinded period) to open-label treatment with everolimus 10mg once daily plus BSC
Period: Blinded Period
Arm/Group | Everolimus + BSC (Throughout Study) | Placebo+BSC (Blinded Period) | Everolimus+BSC (Crossover)
Started | 205 | 97 | 0
Completed (Participants who entered the open-label part of the study) | 26 | 6 | 0
Not Completed | 179 | 91 | 0
Not completed — Adverse Event | 64 | 7 | 0
Not completed — Disease Progression | 89 | 75 | 0
Not completed — Withdrawal by Subject | 19 | 6 | 0
Not completed — Protocol deviation | 2 | 1 | 0
Not completed — Death | 5 | 2 | 0
Period: Open-label Period
Arm/Group | Everolimus + BSC (Throughout Study) | Placebo+BSC (Blinded Period) | Everolimus+BSC (Crossover)
Started | 26 | 0 | 6
Completed | 0 | 0 | 0
Not Completed | 26 | 0 | 6
Not completed — Disease progression | 13 | 0 | 2
Not completed — Administrative problems | 5 | 0 | 2
Not completed — Adverse Event | 5 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Protocol deviation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Everolimus + BSC: Participants received everolimus 10 mg once daily BSC throughout the study
- Placebo+BSC: Participants received matching placebo once daily plus BSC during the blinded period. Participants were allowed to crossover to treatment with everolimus 10mg once daily plus BSC during the open-label period
- Total: Total of all reporting groups
Arm/Group | Everolimus + BSC | Placebo+BSC | Total
Number analyzed (Participants) | 205 | 97 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] — Age continuous at Baseline: Blinded Period
  years | 62.9 (11.70) | 59.4 (12.89) | 61.7 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender at Baseline: Blinded period
  Participants
    Female | 116 | 44 | 160
    Male | 89 | 53 | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race at Baseline: Blinded-period
  Participants
    Caucasian | 162 | 68 | 230
    Asian | 32 | 18 | 50
    Black | 6 | 9 | 15
    Other | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Probability of Participants Remaining Event-Free in Progression-Free Survival (PFS) Based on Central Radiology Assessment
Description: PFS is defined as the time from randomization to the date of the first documented tumor progression or death from any cause, whichever comes first.
  Progression was defined using modified RECIST 1.0 and as per central radiology assessment as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. Progression was assessed by cat scan (CT) and/or magnetic resonance imaging (MRI).
  For participants who had not progressed or died at the analysis cut-off date, PFS was censored at the date of the last adequate tumor evaluation date. An adequate tumour assessment is a tumour assessment with an overall response other than unknown.
  The percentage event-free probability estimate is the estimated probability that a patient will remain event-free in PFS up to the specified time point.
Time Frame: From date of randomization to progression or death, whichever comes first, assessed up to 27 months
Population: The full analysis set (FAS) consists of all randomized patients. Following the intent-to-treat principle, patients were analyzed according to the treatment arm and stratification factors they were assigned to at randomization.
Measure: Number (95% Confidence Interval); unit: Percent event-free probability in PFS
Groups:
- Placebo + BSC: Participants received matching placebo once daily plus BSC during the blinded period. Participants were allowed to crossover to treatment with everolimus 10mg once daily plus BSC during the open-label period
Arm/Group | Everolimus + BSC | Placebo + BSC
Number analyzed (Participants) | 205 | 97
Percent event-free probability in PFS
  2 months | 90.1 [84.8 to 93.5] | 74.6 [64.3 to 82.4]
  4 months | 81.2 [74.9 to 86.2] | 49.1 [38.1 to 59.2]
  6 months | 72.1 [65.0 to 78.0] | 40.1 [29.5 to 50.5]
  8 months | 62.4 [54.8 to 69.1] | 35.8 [25.4 to 46.2]
  10 months | 51.7 [44.0 to 59.0] | 31.3 [21.3 to 41.7]
  12 months | 44.4 [36.7 to 51.8] | 28.1 [18.5 to 38.6]
  15 months | 40.1 [32.5 to 47.6] | 26.4 [16.9 to 36.8]
  18 months | 31.8 [24.1 to 39.8] | 24.4 [15.0 to 34.9]
  21 months | 27.6 [19.0 to 36.8] | 17.4 [9.0 to 28.2]
  24 months | 22.0 [13.0 to 32.5] | 17.4 [9.0 to 28.2]
  27 months | NA [NA to NA] — Not estimable due to the low number of events | 17.4 [9.0 to 28.2]
Statistical Analysis 1: Comparison: Everolimus + BSC vs Placebo + BSC; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.35 to 0.67]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to date of death due to any cause. If a death had not been observed by the date of analysis cut-off, then OS was censored at the date of last contact. All participants randomized to placebo arm who crossed over to everolimus were censored.
Time Frame: From date of randomization to date of death, assessed up to approximately 8 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + BSC | Placebo + BSC
Number analyzed (Participants) | 205 | 97
Months | 43.1 [36.27 to 54.24] | 41.76 [23.46 to 53.75]
Statistical Analysis 1: Comparison: Everolimus + BSC vs Placebo + BSC; Test type: Superiority or Other; p = 0.259, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.66 to 1.24]

3. Secondary Outcome: Overall Response Rate (ORR) as Per Modified RECIST 1.0 According to Central Evaluation
Description: ORR is defined as the proportion of patients with best overall response (BOR) of complete response (CR) or partial response (PR), according to central evaluation and as per modified RECIST 1.0.
  CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters.
Time Frame: From randomization until end of treatment, assessed up to approximately 2.5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + BSC | Placebo + BSC
Number analyzed (Participants) | 205 | 97
Percentage of participants | 2.0 [0.5 to 4.9] | 1.0 [0.0 to 5.6]

4. Secondary Outcome: Disease Control Rate (DCR) Based on Modified RECIST 1.0 and as Per Central Radiology Assessment
Description: DCR is defined as the proportion of subjects with best overall response of CR or PR or stable disease based on modified RECIST 1.0 and as per central radiology assessment.
  CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters.
  Stable disease: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression.
Time Frame: From randomization until end of treatment, assessed up to approximately 2.5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + BSC | Placebo + BSC
Number analyzed (Participants) | 205 | 97
Percentage of participants | 82.4 [76.5 to 87.4] | 64.9 [54.6 to 74.4]

5. Secondary Outcome: Time to Definitive Deterioration in Functional Assessment of Cancer Therapy - General (FACT-G) Questionnaire Total Score
Description: FACT-G is a self-assessed health-related quality of life questionnaire. The questionnaire is comprised of 27 questions examining physical, social/family, emotional, and functional well-being. Participants responded to the items on a five-point scale, ranging from 0: "Not at all" to 4: "Very much." The total score ranges from 0 to 108, with higher scores indicating a better patient-reported outcome/quality of life.
  Definitive deterioration is defined as a decrease in the total score by at least 7 points compared to baseline with no further improvement.
  Death was considered as worsening of the FACT-G total score if it occurred close to the last available assessment, where "close" was defined as twice the planned period between two assessments. Patients without definitive worsening prior to analysis cut-off or prior to start of another anticancer therapy were censored at the date of their last assessment.
Time Frame: From randomization to definitive deterioration of FACT-G total score, assessed up to approximately 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + BSC | Placebo + BSC
Number analyzed (Participants) | 205 | 97
Months | 13.01 [9.33 to 24.80] | 9.23 [5.52 to 28.62]
Statistical Analysis 1: Comparison: Everolimus + BSC vs Placebo + BSC; Test type: Superiority or Other; p = 0.073, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.50 to 1.10]

6. Secondary Outcome: Change From Baseline in Chromogranin A (CgA) Levels
Description: CgA is a potential biomarker for tumor response. Blood samples were collected for assessment of CgA levels. Change from Baseline at a particular visit was calculated as the CgA level at that visit minus Baseline.
Time Frame: From baseline (every 4 weeks) up to 116 weeks
Population: The full analysis set (FAS) consists of all randomized patients. Following the intent-to-treat principle, patients were analyzed according to the treatment arm and stratification factors they were assigned to at randomization. Number analyzed signified number of participants with available data for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: microgram/liter (ug/L)
Arm/Group | Everolimus + BSC | Placebo + BSC
Number analyzed (Participants) | 205 | 97
microgram/liter (ug/L)
  Week 4: number analyzed (Participants) | 164 | 90
  Week 4 | 434.8 (2306.70) | 1154.3 (9083.39)
  Week 8: number analyzed (Participants) | 156 | 88
  Week 8 | 162.3 (2550.65) | 2697.6 (19956.90)
  Week 12: number analyzed (Participants) | 143 | 75
  Week 12 | 396.7 (2401.78) | 1176.0 (3322.13)
  Week 16: number analyzed (Participants) | 141 | 62
  Week 16 | 263.5 (2946.76) | 1450.4 (4825.78)
  Week 20: number analyzed (Participants) | 131 | 51
  Week 20 | 162.1 (2464.47) | 3640.1 (12653.42)
  Week 24: number analyzed (Participants) | 119 | 39
  Week 24 | 253.2 (3487.27) | 1783.9 (5399.98)
  Week 28: number analyzed (Participants) | 112 | 35
  Week 28 | 587.2 (4861.35) | 1350.3 (5701.70)
  Week 32: number analyzed (Participants) | 109 | 31
  Week 32 | 508.5 (6102.61) | 2000.7 (6362.83)
  Week 36: number analyzed (Participants) | 97 | 26
  Week 36 | 94.7 (4905.17) | 180.9 (383.93)
  Week 40: number analyzed (Participants) | 87 | 24
  Week 40 | 511.4 (6180.67) | 207.6 (403.30)
  Week 44: number analyzed (Participants) | 86 | 23
  Week 44 | 552.8 (4173.44) | 140.6 (328.02)
  Week 48: number analyzed (Participants) | 77 | 23
  Week 48 | 1326.2 (8718.92) | 129.0 (326.69)
  Week 52: number analyzed (Participants) | 70 | 24
  Week 52 | 1196.2 (7737.76) | 124.2 (452.38)
  Week 56: number analyzed (Participants) | 60 | 21
  Week 56 | 1920.6 (11250.07) | 134.9 (346.33)
  Week 60: number analyzed (Participants) | 60 | 19
  Week 60 | 1722.0 (13155.03) | 120.9 (415.73)
  Week 64: number analyzed (Participants) | 59 | 19
  Week 64 | 3811.0 (26656.45) | 141.6 (281.38)
  Week 68: number analyzed (Participants) | 56 | 17
  Week 68 | 1413.3 (9588.68) | 222.6 (333.93)
  Week 72: number analyzed (Participants) | 53 | 17
  Week 72 | 239.5 (2318.79) | 233.7 (400.43)
  Week 76: number analyzed (Participants) | 51 | 16
  Week 76 | 3256.5 (19395.40) | 210.9 (522.62)
  Week 80: number analyzed (Participants) | 49 | 15
  Week 80 | 5421.0 (32471.22) | 286.3 (425.45)
  Week 84: number analyzed (Participants) | 45 | 14
  Week 84 | 4379.9 (28302.84) | 175.4 (575.98)
  Week 88: number analyzed (Participants) | 36 | 11
  Week 88 | 571.2 (2694.44) | -9.4 (473.66)
  Week 92: number analyzed (Participants) | 30 | 10
  Week 92 | 765.5 (2913.15) | 63.7 (477.53)
  Week 96: number analyzed (Participants) | 24 | 10
  Week 96 | 984.6 (3379.28) | 146.5 (468.24)
  Week 100: number analyzed (Participants) | 22 | 6
  Week 100 | 935.3 (2961.60) | -12.7 (399.25)
  Week 104: number analyzed (Participants) | 15 | 6
  Week 104 | 1466.4 (4257.03) | -21.7 (285.99)
  Week 108: number analyzed (Participants) | 12 | 6
  Week 108 | 2245.8 (6077.99) | 215.9 (293.87)
  Week 112: number analyzed (Participants) | 12 | 4
  Week 112 | 2817.0 (7786.28) | 514.5 (661.80)
  Week 116: number analyzed (Participants) | 6 | 4
  Week 116 | 2951.8 (6745.06) | 99.6 (92.91)

7. Secondary Outcome: Change From Baseline in Neuron Specific Enolase (NSE) Levels
Description: NSE is a potential biomarker for tumor response. Blood samples were collected for assessment of NSE levels. Change from Baseline at a particular visit was calculated as the NSE level at that visit minus Baseline.
Time Frame: From baseline (every 4 weeks) up to Week 116
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: microgram/liter (ug/L)
Arm/Group | Everolimus + BSC | Placebo + BSC
Number analyzed (Participants) | 205 | 97
microgram/liter (ug/L)
  Week 4: number analyzed (Participants) | 158 | 89
  Week 4 | 0.1 (5.21) | -2.2 (39.87)
  Week 8: number analyzed (Participants) | 151 | 85
  Week 8 | 0.3 (8.71) | -4.2 (36.71)
  Week 12: number analyzed (Participants) | 139 | 74
  Week 12 | -0.3 (8.37) | 15.5 (163.75)
  Week 16: number analyzed (Participants) | 135 | 62
  Week 16 | 2.0 (8.34) | 4.1 (19.44)
  Week 20: number analyzed (Participants) | 128 | 50
  Week 20 | 0.8 (6.21) | 5.3 (18.26)
  Week 24: number analyzed (Participants) | 117 | 39
  Week 24 | 1.7 (8.99) | 6.7 (23.47)
  Week 28: number analyzed (Participants) | 110 | 35
  Week 28 | 1.1 (6.37) | 0.4 (9.16)
  Week 32: number analyzed (Participants) | 106 | 31
  Week 32 | 1.5 (14.24) | 3.1 (8.96)
  Week 36: number analyzed (Participants) | 96 | 27
  Week 36 | 2.0 (15.11) | 2.0 (5.90)
  Week 40: number analyzed (Participants) | 86 | 24
  Week 40 | 1.2 (6.48) | 1.2 (4.49)
  Week 44: number analyzed (Participants) | 87 | 23
  Week 44 | 0.8 (5.10) | 1.2 (4.46)
  Week 48: number analyzed (Participants) | 74 | 23
  Week 48 | 2.0 (9.20) | 0.6 (4.06)
  Week 52: number analyzed (Participants) | 71 | 23
  Week 52 | 1.5 (5.82) | 0.7 (4.19)
  Week 56: number analyzed (Participants) | 60 | 21
  Week 56 | 3.6 (18.56) | 0.9 (5.89)
  Week 60: number analyzed (Participants) | 63 | 20
  Week 60 | 2.4 (8.19) | 0.1 (3.35)
  Week 64: number analyzed (Participants) | 58 | 18
  Week 64 | 4.4 (23.22) | 0.9 (3.80)
  Week 68: number analyzed (Participants) | 58 | 18
  Week 68 | 1.1 (4.68) | 1.9 (4.48)
  Week 72: number analyzed (Participants) | 53 | 18
  Week 72 | 1.6 (4.46) | 0.7 (3.91)
  Week 76: number analyzed (Participants) | 52 | 16
  Week 76 | 1.7 (5.11) | 0.6 (3.89)
  Week 80: number analyzed (Participants) | 51 | 13
  Week 80 | 2.9 (10.15) | 0.7 (2.83)
  Week 84: number analyzed (Participants) | 41 | 14
  Week 84 | 8.0 (33.13) | 0.1 (3.47)
  Week 88: number analyzed (Participants) | 37 | 11
  Week 88 | 2.2 (3.89) | 0.6 (2.47)
  Week 92: number analyzed (Participants) | 29 | 10
  Week 92 | 4.0 (7.24) | 0.1 (3.79)
  Week 96: number analyzed (Participants) | 23 | 10
  Week 96 | 4.3 (5.96) | 0.0 (2.99)
  Week 100: number analyzed (Participants) | 22 | 5
  Week 100 | 1.8 (3.79) | -0.2 (5.10)
  Week 104: number analyzed (Participants) | 15 | 6
  Week 104 | 2.9 (4.11) | -1.7 (4.76)
  Week 108: number analyzed (Participants) | 12 | 6
  Week 108 | 5.5 (13.48) | -0.5 (4.33)
  Week 112: number analyzed (Participants) | 11 | 3
  Week 112 | 2.8 (5.72) | -3.2 (3.30)
  Week 116: number analyzed (Participants) | 6 | 4
  Week 116 | 10.6 (14.92) | 0.2 (4.17)

8. Secondary Outcome: Time to Definitive Deterioration in World Health Organization (WHO) Performance Status (PS) Change
Description: WHO PS is a scale rated from 0 (fully active) to 5 (death) by a healthcare professional to assess the overall status of a patient: a lower score represents a higher ability to perform daily tasks. Deterioration is defined as an increase of at least one point compared to baseline. Deterioration is considered definitive if no improvements in the WHO PS status is observed at a subsequent time of measurement during the treatment period following the time point where the deterioration is observed. Death was considered as worsening of the WHO PS if it occurred close to the last available assessment, where "close" was defined as twice the planned period between two assessments. Patients without definitive worsening prior to analysis cut-off or prior to start of another anticancer therapy were censored at the date of their last assessment.
Time Frame: From randomization to definitive deterioration of WHO performance status, assessed up to approximately 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + BSC | Placebo + BSC
Number analyzed (Participants) | 205 | 97
Months | 24.08 [17.05 to NA] — NA. Not evaluable due to the low number of participants with an event of interest. | 24.15 [8.31 to NA] — NA. Not evaluable due to the low number of participants with an event of interest.
Statistical Analysis 1: Comparison: Everolimus + BSC vs Placebo + BSC; Test type: Superiority or Other; p = 0.539, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.65 to 1.61]

9. Secondary Outcome: Pharmacokinetics (PK): Predose Concentration (Cmin) of Everolimus at Day 29
Description: A pre-dose blood sample at day 29 was collected to determine the exposure of everolimus at the steady-state pre-dose concentration (Cmin). Cmin is provided for participants randomized to everolimus+BSC who received 10mg of everolimus daily and also for participants randomized to everolimus+BSC who received 5mg of everolimus daily which was required for a number of participants in the study experiencing adverse events requiring dose modifications
Time Frame: Pre-dose at Day 29.
Population: All patients who received at least one dose of the study drug with evaluable blood samples for this endpoint.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Everolimus + BSC
Number analyzed (Participants) | 48
nanogram/milliliter (ng/mL)
  10mg daily dose | 16.382 (13.2767)
  5mg daily dose: number analyzed (Participants) | 3
  5mg daily dose | 4.700 (3.8396)

10. Post Hoc Outcome: All Collected Deaths
Description: Deaths on-treatment were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of approximately 8 years.
  Total Deaths were collected from first dose of study treatment until end of post-treatment survival follow, up to maximum duration of approximately 8 years.
Time Frame: On-treatment deaths: up to approximately 8 years. All deaths: up to approximately 8 years
Population: The safety set consists of all participants who received at least one dose of the study drug and had at least one post-baseline safety evaluation. Participants were analyzed according to treatment actually received: One participant randomized to everolimus arm received only placebo and therefore, appears in the placebo arm in the safety set
Measure: Number; unit: Participants
Groups:
- Everolimus + BSC (Throughout the Study): Participants received everolimus 10 mg once daily BSC throughout the study
- Everolimus +BSC (Crossover): Participants who crossed over from placebo arm (blinded period) to open-label treatment with everolimus 10mg once daily plus BSC
- Everolimus+BSC (All): All participants who received everolimus 10 mg once daily plus BSC (including those who received everolimus+BSC from start to end of the study and those who received everolimus+BSC after crossover)
- Placebo + BSC (Blinded Period): Participants received matching placebo once daily plus BSC during the blinded period
Arm/Group | Everolimus + BSC (Throughout the Study) | Everolimus +BSC (Crossover) | Everolimus+BSC (All) | Placebo + BSC (Blinded Period)
Number analyzed (Participants) | 202 | 6 | 208 | 98
Participants
  On-treatment deaths | 10 | 0 | 10 | 5
  Total deaths | 126 | 1 | 127 | 57

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were collected from date of first dose of study treatment until end of study treatment plus 30 days post treatment, assessed up to a maximum duration of approximately 8 years
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment. The safety set consists of all participants who received at least one dose of the study drug and had at least one post-baseline safety evaluation. Participants were analyzed according to treatment actually received: One participant randomized to everolimus arm received only placebo and therefore, appears in the placebo arm in the safety set
Groups:
- Everolimus+BSC (Throughout Study): Participants received everolimus 10 mg once daily plus BSC throughout the study
- Placebo+BSC (Blinded Period): Participants received matching placebo once daily plus best supportive care (BSC) during the blinded period.
Arm/Group | Everolimus+BSC (Throughout Study) | Everolimus +BSC (Crossover) | Everolimus+BSC (All) | Placebo+BSC (Blinded Period)
All-Cause Mortality (participants affected / at risk) | 10/202 | 0/6 | 10/208 | 5/98
Serious Adverse Events (participants affected / at risk) | 93/202 | 1/6 | 94/208 | 21/98
Other Adverse Events (participants affected / at risk) | 197/202 | 6/6 | 203/208 | 81/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus+BSC (Throughout Study) (N=202) | Everolimus +BSC (Crossover) (N=6) | Everolimus+BSC (All) (N=208) | Placebo+BSC (Blinded Period) (N=98)
Anaemia (Blood and lymphatic system disorders) | 7 | 0 | 7 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 0 | 3 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 0 | 3 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 13 | 1 | 14 | 4
Ascites (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 0 | 10 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Gastrointestinal oedema (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0 | 3 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Jejunal perforation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 3 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatic necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 6 | 1 | 7 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 5 | 2
Asthenia (General disorders) | 6 | 0 | 6 | 0
Chest discomfort (General disorders) | 1 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 7 | 0 | 7 | 0
General physical health deterioration (General disorders) | 1 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 2 | 0 | 2 | 1
Organ failure (General disorders) | 1 | 0 | 1 | 0
Performance status decreased (General disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 11 | 0 | 11 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 0 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 0 | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 2 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 0 | 2 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Contrast media allergy (Immune system disorders) | 1 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 1 | 0
Incision site cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Infection (Infections and infestations) | 2 | 0 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 2 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 7 | 0 | 7 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 2 | 0
Salmonellosis (Infections and infestations) | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Septic shock (Infections and infestations) | 2 | 0 | 2 | 0
Skin infection (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 0 | 4 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 1 | 0
Viral myocarditis (Infections and infestations) | 1 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 0 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 2 | 0
Gastrointestinal stoma output decreased (Investigations) | 1 | 0 | 1 | 0
Troponin increased (Investigations) | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 3 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1
Stress (Psychiatric disorders) | 1 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 0 | 4 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus+BSC (Throughout Study) (N=202) | Everolimus +BSC (Crossover) (N=6) | Everolimus+BSC (All) (N=208) | Placebo+BSC (Blinded Period) (N=98)
Anaemia (Blood and lymphatic system disorders) | 47 | 0 | 47 | 9
Deafness (Ear and labyrinth disorders) | 1 | 1 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 2 | 5 | 2
Carcinoid syndrome (Endocrine disorders) | 1 | 1 | 2 | 0
Blindness (Eye disorders) | 0 | 1 | 1 | 0
Dry eye (Eye disorders) | 4 | 1 | 5 | 0
Eye pain (Eye disorders) | 1 | 1 | 2 | 0
Visual impairment (Eye disorders) | 0 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 8
Abdominal pain (Gastrointestinal disorders) | 38 | 1 | 39 | 17
Abdominal pain upper (Gastrointestinal disorders) | 21 | 0 | 21 | 11
Aphthous ulcer (Gastrointestinal disorders) | 8 | 3 | 11 | 2
Constipation (Gastrointestinal disorders) | 25 | 2 | 27 | 19
Diarrhoea (Gastrointestinal disorders) | 88 | 3 | 91 | 30
Dry mouth (Gastrointestinal disorders) | 18 | 0 | 18 | 5
Dyspepsia (Gastrointestinal disorders) | 11 | 1 | 12 | 5
Flatulence (Gastrointestinal disorders) | 7 | 1 | 8 | 6
Mouth ulceration (Gastrointestinal disorders) | 18 | 0 | 18 | 1
Nausea (Gastrointestinal disorders) | 58 | 0 | 58 | 16
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 113 | 2 | 115 | 19
Tongue ulceration (Gastrointestinal disorders) | 2 | 1 | 3 | 0
Toothache (Gastrointestinal disorders) | 11 | 2 | 13 | 3
Vomiting (Gastrointestinal disorders) | 33 | 0 | 33 | 10
Asthenia (General disorders) | 46 | 0 | 46 | 9
Chills (General disorders) | 6 | 1 | 7 | 1
Fatigue (General disorders) | 76 | 2 | 78 | 36
Oedema peripheral (General disorders) | 81 | 1 | 82 | 5
Peripheral swelling (General disorders) | 11 | 0 | 11 | 2
Pyrexia (General disorders) | 49 | 2 | 51 | 9
Hypersensitivity (Immune system disorders) | 1 | 1 | 2 | 0
Bronchitis (Infections and infestations) | 8 | 2 | 10 | 2
Cystitis (Infections and infestations) | 7 | 1 | 8 | 1
Gastrointestinal viral infection (Infections and infestations) | 1 | 1 | 2 | 0
Influenza (Infections and infestations) | 9 | 2 | 11 | 1
Nasopharyngitis (Infections and infestations) | 22 | 2 | 24 | 4
Pneumonia (Infections and infestations) | 18 | 0 | 18 | 0
Pulpitis dental (Infections and infestations) | 0 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 4 | 1 | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 18 | 1 | 19 | 6
Urinary tract infection (Infections and infestations) | 23 | 1 | 24 | 6
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 4 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 12 | 0 | 12 | 2
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 3 | 5
Blood creatinine increased (Investigations) | 11 | 1 | 12 | 1
Blood urea (Investigations) | 0 | 1 | 1 | 0
Blood uric acid (Investigations) | 0 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 9 | 1 | 10 | 2
Weight decreased (Investigations) | 51 | 2 | 53 | 11
Decreased appetite (Metabolism and nutrition disorders) | 53 | 1 | 54 | 17
Hypercholesterolaemia (Metabolism and nutrition disorders) | 16 | 1 | 17 | 2
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 24 | 1 | 25 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 12 | 1 | 13 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 3 | 24 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 1 | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 0 | 31 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 0 | 34 | 14
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 0 | 15 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 0 | 19 | 5
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 11 | 0 | 11 | 5
Dysgeusia (Nervous system disorders) | 26 | 1 | 27 | 3
Headache (Nervous system disorders) | 27 | 1 | 28 | 15
Paraesthesia (Nervous system disorders) | 5 | 2 | 7 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 2 | 1
Taste disorder (Nervous system disorders) | 13 | 1 | 14 | 1
Anxiety (Psychiatric disorders) | 9 | 1 | 10 | 1
Insomnia (Psychiatric disorders) | 20 | 0 | 20 | 8
Dysuria (Renal and urinary disorders) | 8 | 0 | 8 | 5
Haematuria (Renal and urinary disorders) | 11 | 1 | 12 | 4
Proteinuria (Renal and urinary disorders) | 18 | 0 | 18 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 63 | 1 | 64 | 20
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 7 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 42 | 0 | 42 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28 | 2 | 30 | 3
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 1 | 14 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 0 | 12 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 30 | 0 | 30 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 20 | 0 | 20 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 0 | 18 | 2
Eczema (Skin and subcutaneous tissue disorders) | 6 | 1 | 7 | 0
Erythema (Skin and subcutaneous tissue disorders) | 11 | 0 | 11 | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 37 | 2 | 39 | 9
Rash (Skin and subcutaneous tissue disorders) | 62 | 3 | 65 | 9
Hypertension (Vascular disorders) | 28 | 1 | 29 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in the clinical trial